CLINICAL TRIAL: NCT03696524
Title: Tunneled Pleural Catheters for Refractory Effusions Attributed to Congestive Heart Failure (TREAT-CHF) Trial
Acronym: TREAT-CHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Scott S. Oh, DO, FCCP, DAABIP, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-000400
Record Dates: First submitted 2018-09-11; First posted 2018-10-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pleural Effusions, Chronic; Congestive Heart Failure; Shortness of Breath
Keywords: congestive heart failure; pleural effusion; shortness of breath; tunneled pleural catheter; thoracentesis
MeSH Terms: conditions — Pleural Effusion; Bronchiolitis Obliterans Syndrome; Heart Failure; Dyspnea

STUDY DESIGN:
Intervention Model Description: There will be an intervention group (receiving the tunneled pleural catheter) and a usual care group.
Who Masked: Outcomes Assessor
Masking Description: The subjects and providers will not be blinded, since it will be apparent which patients received a pleurx catheter. Outcomes measured by survey and chart review will be scored and analyzed in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group will receive placement of a tunneled pleural catheter to drain their recurrent, chronic, and symptomatic pleural effusion in addition to their usual medication therapy.
  Interventions: Device: tunneled pleural catheter
- Usual Care (No Intervention): The control group will continue with medical therapy by their referring physician and serial thoracenteses when clinically appropriate.

INTERVENTIONS:
Device: tunneled pleural catheter — Placement of a tunneled pleural catheter through the chest wall into the pleural space to drain the patient's chronic pleural effusion. The catheter is an indwelling device that will be drained from home three times per week by nursing care, the patient, or patient's family.
  Other Names: pleurx catheter placement
  Arms: Intervention Group

SUMMARY:
Congestive heart disease (CHF) can frequently cause transudative pleural effusions, some of which do not completely resolve with diuretics alone. These effusions can cause significant morbidity, leading to ongoing dyspnea and hypoxia, resulting in additional office and hospital visits. TREAT-CHF is a randomized trial studying tunneled pleural catheter (TPC) versus standard medical management for the treatment recurrent symptomatic pleural effusions secondary to CHF that are refractory to maximal medical therapy. TREAT-CHF will study whether the addition of a TPC can improve quality of life and minimize health care utilization over the one year following insertion.

DETAILED DESCRIPTION:
TREAT-CHF is a randomized trial studying tunneled pleural catheter (TPC) versus standard medical management for the treatment recurrent symptomatic pleural effusions secondary to CHF that are refractory to maximal medical therapy. All trial participants will be adults with congestive heart failure (CHF) already managed with maximal medical therapy, as determined by their cardiologist or primary physician. Patients will demonstrate recurrent transudative or pseudoexudative pleural effusions caused solely by CHF that have not been controlled with medical therapy alone. Included patients must also show documented subjective symptomatic relief with thoracentesis.

Patients will be randomized to the intervention group or control group. The intervention group will receive a tunneled pleural catheter (TPC) in addition to their current medical treatment. The control group will continue with medical therapy by their referring physician and serial thoracenteses when clinically appropriate. Patients will then be followed over the course of once year after enrollment. The TPC will be drained daily for symptomatic relief. Several outcomes, including quality of life based on periodic self-survey and healthcare utilization determined by chart review (emergency room visits and hospital stays), will be studied. Adverse outcomes of TPC insertion and sequelae of frequent pleural space drainage will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age at enrollment
2. Able to give consent
3. Documented heart failure defined by echocardiography demonstrating depressed left ventricular ejection fraction and/or left ventricular diastolic dysfunction
4. Recurrent and symptomatic pleural effusions refractory to medical management
5. Maximal medical management will be determined by the referring provider a. This should include use of at least three of the classes of medications that are standard of care for heart failure: i. Angiotensin converting enzyme inhibitor or angiotensin receptor blockers ii. Beta blockers iii. Loop diuretics iv. Potassium-sparing diuretics b. If the patient is not on at least three drugs from the above classes, documentation of drug intolerance must be present
6. Documented subjective symptomatic relief after thoracentesis and drainage of the pleural space
7. Pleural fluid clinically determined to be due only to CHF
8. Pleural fluid analysis consistent with transudate or pseudoexudate a. Transudate: defined by Light's criteria, all of the following must occur, i. Pleural:serum lactate dehydrogenase (LDH) < 0.6 ii. Pleural LDH < 2/3 x upper limit of normal of serum LDH iii. Pleural:serum protein < 0.5 b. Pseudoexudate: defined by all of the following, i. Pleural:serum LDH > 0.6 but < 1 ii. Pleural:serum protein < 0.5 iii. Serum-pleural protein gradient > 3.2 and/or serum-pleural albumin gradient > 1.2
9. Anticipated outpatient management

Exclusion Criteria:

1. Imminent death within 1 month
2. Heart transplant candidate
3. Lone right sided heart failure with normal left sided cardiac function
4. Active malignancy
5. Active pulmonary infection
6. Alternate etiology for pleural effusion origin
7. On hemodialysis during enrollment
8. Exudative pleural effusion, defined as any effusion that dose not meet criteria for transudate or pseudoexudate
9. Contraindication for TPC insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life scores from baseline as measured by the Minnesota Living with Heart Failure Questionnaire | Change from baseline at 3 time points over the year of follow up (3, 6, and 12 months)
  Quality of life will be measured by the Minnesota Living with Heart Failure Questionnaire at four time points
Incidence of hospitalizations and emergency room encounters | 1 year post-enrollment
  Measurement of all significant health care visits, including hospitalizations and emergency room encounters

SECONDARY OUTCOMES:
All cause mortality | 1 year post-enrollment
  All cause mortality
New York Heath Association (NYHA) functional class | Change from baseline at 3 time points over the year of follow up (3, 6, and 12 months)
  NYHA functional class: I, III, III, or IV
Incidence of pleural procedures | 1 year post-enrollment
  By convention, the intervention group will have one pleural procedure (TPC placement). Any additional thoracenteses, video-assisted thoracoscopic surgery, or chest tubes on either side of the chest will be documented for both groups. Removal of or manipulation of TPC will not be recorded as an additional pleural procedure.
Incidence of pleural space or chest wall infection | 1 year post-enrollment
  Pleural space infection is defined as a positive pleural fluid culture. Chest wall infection will be defined clinically, based on the presence of cellulitis surrounding the catheter or catheter tract, or pus draining from the catheter insertion site.
Incidence of hemothorax | 1 year post-enrollment
  Hemothorax is defined as a pleural hematocrit or red blood cell count (RBC) exceeding 50% that of the serum hematocrit or RBC count.
Incidence of trapped lung, loculated pleural effusion, and pneumothorax | 1 year post-enrollment
  Trapped lung is defined as a lung that does not expand after pleural fluid drainage leaving a pneumothorax ex-vacuo or hydropneumothorax. Pneumothorax and loculated pleural effusion will be determined based on classic imaging characteristics.
Incidence of pleurodesis | 1 year post-enrollment
  Incidence of pleurodesis over the one year after enrollment will be measured. Pleurodesis is defined as apposition of the parietal and visceral pleural such: (i) that the subject drains less than 10cc on three serial drainages, (ii) there is resolution of the pleural effusion on both chest x-ray (CXR) and chest ultrasound, (iii) the TPC is removed, and (iv) the pleural effusion does not accumulate after TPC removal as evidence by CXR and chest ultrasound.
Time to pleurodesis among those who achieved pleurodesis | 1 year post-enrollment
  The number of days from enrollment (control group) or TPC placement (intervention group) to pleurodesis among those who achieved pleurodesis will be recorded. Pleurodesis is defined as apposition of the parietal and visceral pleural such: (i) that the subject drains less than 10cc on three serial drainages, (ii) there is resolution of the pleural effusion on both chest x-ray (CXR) and chest ultrasound, (iii) the TPC is removed, and (iv) the pleural effusion does not accumulate after TPC removal as evidence by CXR and chest ultrasound.
Change from baseline serum albumin | Change from baseline at 3 time points over the year of follow up (3, 6, and 12 months)
  serum albumin levels
Change from baseline serum creatinine | Change from baseline at 3 time points over the year of follow up (3, 6, and 12 months)
  serum creatinine levels
Rate of hemodialysis initiation | 1 year post-enrollment
  We will record patients who develop worsening renal failure, necessitating initiation of hemodialysis

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freeman RK, Ascioti AJ, Dake M, Mahidhara RS. A propensity-matched comparison of pleurodesis or tunneled pleural catheter for heart failure patients with recurrent pleural effusion. Ann Thorac Surg. 2014 Jun;97(6):1872-6; discussion 1876-7. doi: 10.1016/j.athoracsur.2014.02.027. Epub 2014 Apr 14. PMID 24726601
- [Background] Roberts ME, Neville E, Berrisford RG, Antunes G, Ali NJ; BTS Pleural Disease Guideline Group. Management of a malignant pleural effusion: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii32-40. doi: 10.1136/thx.2010.136994. No abstract available. PMID 20696691
- [Background] Light RW, Macgregor MI, Luchsinger PC, Ball WC Jr. Pleural effusions: the diagnostic separation of transudates and exudates. Ann Intern Med. 1972 Oct;77(4):507-13. doi: 10.7326/0003-4819-77-4-507. No abstract available. PMID 4642731
- [Background] Davies HE, Mishra EK, Kahan BC, Wrightson JM, Stanton AE, Guhan A, Davies CW, Grayez J, Harrison R, Prasad A, Crosthwaite N, Lee YC, Davies RJ, Miller RF, Rahman NM. Effect of an indwelling pleural catheter vs chest tube and talc pleurodesis for relieving dyspnea in patients with malignant pleural effusion: the TIME2 randomized controlled trial. JAMA. 2012 Jun 13;307(22):2383-9. doi: 10.1001/jama.2012.5535. PMID 22610520
- [Background] Light RW. Clinical practice. Pleural effusion. N Engl J Med. 2002 Jun 20;346(25):1971-7. doi: 10.1056/NEJMcp010731. No abstract available. PMID 12075059
- [Background] Porcel JM, Light RW. Diagnostic approach to pleural effusion in adults. Am Fam Physician. 2006 Apr 1;73(7):1211-20. PMID 16623208
- [Background] EDWARDS JE, RACE GA, SCHEIFLEY CH. Hydrothorax in congestive heart failure. Am J Med. 1957 Jan;22(1):83-9. doi: 10.1016/0002-9343(57)90339-x. No abstract available. PMID 13381740
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Majid A, Kheir F, Fashjian M, Chatterji S, Fernandez-Bussy S, Ochoa S, Cheng G, Folch E. Tunneled Pleural Catheter Placement with and without Talc Poudrage for Treatment of Pleural Effusions Due to Congestive Heart Failure. Ann Am Thorac Soc. 2016 Feb;13(2):212-6. doi: 10.1513/AnnalsATS.201507-471BC. PMID 26598967
- [Background] Krishnan M, Cheriyath P, Wert Y, Moritz TA. The Untapped Potential of Tunneled Pleural Catheters. Ann Thorac Surg. 2015 Dec;100(6):2055-7. doi: 10.1016/j.athoracsur.2015.05.086. Epub 2015 Aug 18. PMID 26294344
- [Background] Srour N, Potechin R, Amjadi K. Use of indwelling pleural catheters for cardiogenic pleural effusions. Chest. 2013 Nov;144(5):1603-1608. doi: 10.1378/chest.13-0331. PMID 23807028
- [Background] Chalhoub M, Harris K, Castellano M, Maroun R, Bourjeily G. The use of the PleurX catheter in the management of non-malignant pleural effusions. Chron Respir Dis. 2011;8(3):185-91. doi: 10.1177/1479972311407216. Epub 2011 Jun 2. PMID 21636653
- [Background] Chakko SC, Caldwell SH, Sforza PP. Treatment of congestive heart failure. Its effect on pleural fluid chemistry. Chest. 1989 Apr;95(4):798-802. doi: 10.1378/chest.95.4.798. PMID 2924609
- [Background] Romero-Candeira S, Fernandez C, Martin C, Sanchez-Paya J, Hernandez L. Influence of diuretics on the concentration of proteins and other components of pleural transudates in patients with heart failure. Am J Med. 2001 Jun 15;110(9):681-6. doi: 10.1016/s0002-9343(01)00726-4. PMID 11403751
- [Background] Roth BJ, O'Meara TF, Cragun WH. The serum-effusion albumin gradient in the evaluation of pleural effusions. Chest. 1990 Sep;98(3):546-9. doi: 10.1378/chest.98.3.546. PMID 2152757
- [Background] Bottle A, Goudie R, Bell D, Aylin P, Cowie MR. Use of hospital services by age and comorbidity after an index heart failure admission in England: an observational study. BMJ Open. 2016 Jun 9;6(6):e010669. doi: 10.1136/bmjopen-2015-010669. PMID 27288372
- [Background] Kawano H, Arakawa S, Satoh O, Matsumoto Y, Hayano M, Nakatomi D, Yamasa T, Maemura K. Effect of pimobendan in addition to standard therapy for heart failure on prevention of readmission in elderly patients with severe chronic heart failure. Geriatr Gerontol Int. 2014 Jan;14(1):109-14. doi: 10.1111/ggi.12067. Epub 2013 Apr 15. PMID 23581555
- [Background] Bennett SJ, Oldridge NB, Eckert GJ, Embree JL, Browning S, Hou N, Chui M, Deer M, Murray MD. Comparison of quality of life measures in heart failure. Nurs Res. 2003 Jul-Aug;52(4):207-16. doi: 10.1097/00006199-200307000-00001. PMID 12867777